CLINICAL TRIAL: NCT02698267
Title: An Open-label, Fixed-sequence, Phase 1 Study of the Effect of CYP3A4 Inhibition by Itraconazole on the Pharmacokinetics of BIIB074 in Healthy Subjects
Brief Title: Effect of Itraconazole on the Pharmacokinetics of BIIB074
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 802HV104; 2015-005096-25 (EudraCT Number)
Record Dates: First submitted 2016-02-29; First posted 2016-03-03 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — vixotrigine; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BIIB074 (Experimental): Administered orally on Day 1 and Day 11
  Interventions: Drug: BIIB074; Drug: Itraconazole

INTERVENTIONS:
Drug: BIIB074 — Administered as specified in the treatment arm
  Other Names: CNV1014802
Drug: Itraconazole — 200 mg twice daily [BID] on Day 8 and once daily (QD) from Day 9 to Day 15 inclusive
  Other Names: Sporanox, Onmel

SUMMARY:
The primary objective of the study is to assess the effect of cytochrome P450 (CYP) 3A4 inhibition on the pharmacokinetics (PK) of BIIB074. The secondary objectives of this study are to assess the safety and tolerability of BIIB074 when co-administered with a strong CYP3A4 inhibitor and to assess the effect of CYP3A4 inhibition on the PK of 3 metabolites of BIIB074 (CNV3000497 [M13], CNV2283325 [M14], and CNV2288584 [M16]).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index of 18 to 29 kg/m2, inclusive, with body weight ≥50 kg for males and ≥45 kg for females.
* Male or postmenopausal or surgically sterile females.
* Must be in good health as determined by the Investigator (or designee), based on medical history and screening evaluations.

Key Exclusion Criteria:

* Females of childbearing potential.
* Other unspecified reasons that, in the opinion of the Investigator or Sponsor, make the subject unsuitable for enrollment.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) of BIIB074 | Prior to dosing up to 96 hours post dose
Exposure of BIIB074 as measured by area under the concentration-time curve from time zero to infinity (AUCinf) | Prior to dosing up to 96 hours post dose

SECONDARY OUTCOMES:
Terminal elimination half-life (t1/2) of BIIB074 | 96 hours post dose
Apparent total body clearance (CL/F) of BIIB074 | 96 hours post dose
Apparent volume of distribution (Vd/F) of BIIB074 | 96 hours post dose
Area under the concentration-time curve from time zero to time of the last measurable drug concentration (AUC0-t) of BIIB074 | Prior to dosing up to 96 hours post dose
Time that the maximum observed concentration occurs (Tmax) of BIIB074 | Prior to dosing up to 96 hours post dose
Number of participants experiencing adverse events (AEs) and serious adverse events (SAEs) | Up to 25 days
Number of participants with clinically significant vital sign abnormalities | Up to 25 days
Number of participants with clinically significant 12-lead electrocardiograms (ECGs) abnormalities | Up to 25 days
Number of participants with clinically significant laboratory assessment abnormalities | Up to 25 days
Effect of CYP3A4 inhibition on the Cmax of 3 metabolites of BIIB074 | Prior to dosing up to 96 hours post dose
Effect of CYP3A4 inhibition on the AUCinf of 3 metabolites of BIIB074 | Prior to dosing up to 96 hours post dose
Effect of CYP3A4 inhibition on the AUC0-t of CNV3000497 (M13) | Prior to dosing up to 96 hours post dose
Effect of CYP3A4 inhibition on the AUC0-t of CNV2283325 (M14) | Prior to dosing up to 96 hours post dose
Effect of CYP3A4 inhibition on the AUC0-t of CNV2288584 (M16) | Prior to dosing up to 96 hours post dose
Effect of CYP3A4 inhibition on the Tmax of CNV3000497 (M13) | Prior to dosing up to 96 hours post dose
Effect of CYP3A4 inhibition on the Tmax of CNV2283325 (M14) | Prior to dosing up to 96 hours post dose
Effect of CYP3A4 inhibition on the Tmax of CNV2288584 (M16) | Prior to dosing up to 96 hours post dose
Effect of CYP3A4 inhibition on the t1/2 of CNV3000497 (M13) | Prior to dosing up to 96 hours post dose
Effect of CYP3A4 inhibition on the t1/2 of CNV2283325 (M14) | Prior to dosing up to 96 hours post dose
Effect of CYP3A4 inhibition on the t1/2 of CNV2288584 (M16) | Prior to dosing up to 96 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Leeds, United Kingdom